CLINICAL TRIAL: NCT03964922
Title: Study of the Immunoevasive Mecanisms and Especially Myeloid Suppressive Cells in the Medullar Microenvironment Employed by Myeloid Malignancy (AML and High Risk MDS) When Relapsing After Allogeneic Stem Cell Transplantation
Brief Title: Immunoevasive Tactics Employed by Myeloid Malignancy After Allogeneic Stem Cell Transplantation
Acronym: EVADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-A00842-55
Record Dates: First submitted 2019-05-03; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Relapse Leukemia; Allogeneic Stem Cell Transplantation; Immune Evasion, Tumor
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immune escape mecanims (Experimental): Cohort study with a representative sample of patients
  Interventions: Biological: blood sample; Biological: bone marrow sample

INTERVENTIONS:
Biological: blood sample — 20 ml at inclusion, and 20ml at 1, 3, 6 and 12 months after allo HSCT
Biological: bone marrow sample — 3 ml at inclusion, and 3 ml at 1, 3, 6 and 12 months after allo HSCT

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is still the only treatment available to cure acute myeloid leukemia and high risk myelodysplasia. Allo-HSCT has an anti-tumor effect (called the graft versus leukemia effect= GVL) mediated by donor lymphocytes. This GVL effect is often associated with graft-versus-host disease (GVHD). Several studies have shown that the relapse incidence is lower in patients developing chronic GVHD. These studies confirm the impact of donor immune system on leukemic residual cells. In fact, the relapse incidence increased in patients with no sign of GVHD. The investigators assume that leukemic cells probably use mechanisms to inhibit the allogeneic response. These escape mechanisms to immunosurveillance have been described in other malignancies. Out of context of the allo-HSCT, in acute myeloid leukemias and myelodysplasia, correlations between the severity of the disease and the presence of regulatory T cells (Tregs) or exhausted T cells (PD1 positive) in the bone marrow and in the blood of patients were described at the time of diagnosis or relapse. Myeloid Derived Suppressive Cells (MDSCs) have been described as capable of inducing Tregs and exhausted T cells in the tumor microenvironment.The investigators want to evaluate the role of myeloid suppressive cells in bone marrow after allo HSCT. They hypothesize that their presence in bone marrow and / or blood recipient is correlated to the relapse incidence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myeloid leukemia in complete cytological remission with intermediate or high risk prognosis according to ELN 2017
* Patients with myelodysplasia according to the WHO 2016 definition, with IPSS ≥1.5 and disease status is : stable or in partial response or complete response according to IWG 2006.
* Patients with indication of first allo-HSCT with a matched related or unrelated donor
* Patients receiving non-myeloablative or reduced toxicity conditioning
* Patients affiliated to a social security scheme
* Patients who have received a complete information on the organization of the research and signed his informed consent

Exclusion Criteria:

* Patients with an alternative donor (HLA 5/10 or unit cord blood)
* Patients with another active cancer or a history of cancer diagnosed in the previous 5 years
* Patients with uncontrolled infection at the time of inclusion, or with positive HIV (1 + 2) or HTLV (1 + 2), Hepatitis C or active hepatitis B
* Patients referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Myeloid suppressive cells and relapse incidence | 2 years
  To investigate the relationship between the percentage of myeloid derived suppressive cells (MDSCs) in total leukocytes in peripheral blood and the relapse incidence after allogeneic stem cell transplantation.
  The patients will be grouped according to median MDSC frequency values. Relapse incidence will be compared across the two groups (low and high frequency of MDSC).

SECONDARY OUTCOMES:
Myeloid suppressive cells and the medullar microenvironment (regulatory T cells and mesenchymal stem cells) | 2 years
  To correlate levels of bone marrow MDSC and regulatory T cells (Tregs) and exhausted T cells and the quality of mesenchymal cells in bone marrow.
percentage of myeloid suppressive cells | 2 years
incidence of acute GVHD | 2 years
incidence of chronic GVHD | 2 years

REFERENCES:
- [Background] D'Aveni M, Rossignol J, Coman T, Sivakumaran S, Henderson S, Manzo T, Santos e Sousa P, Bruneau J, Fouquet G, Zavala F, Alegria-Prevot O, Garfa-Traore M, Suarez F, Trebeden-Negre H, Mohty M, Bennett CL, Chakraverty R, Hermine O, Rubio MT. G-CSF mobilizes CD34+ regulatory monocytes that inhibit graft-versus-host disease. Sci Transl Med. 2015 Apr 1;7(281):281ra42. doi: 10.1126/scitranslmed.3010435. PMID 25834108
- [Background] Kumar B, Garcia M, Weng L, Jung X, Murakami JL, Hu X, McDonald T, Lin A, Kumar AR, DiGiusto DL, Stein AS, Pullarkat VA, Hui SK, Carlesso N, Kuo YH, Bhatia R, Marcucci G, Chen CC. Acute myeloid leukemia transforms the bone marrow niche into a leukemia-permissive microenvironment through exosome secretion. Leukemia. 2018 Mar;32(3):575-587. doi: 10.1038/leu.2017.259. Epub 2017 Aug 17. PMID 28816238
- [Background] Nadal E, Garin M, Kaeda J, Apperley J, Lechler R, Dazzi F. Increased frequencies of CD4(+)CD25(high) T(regs) correlate with disease relapse after allogeneic stem cell transplantation for chronic myeloid leukemia. Leukemia. 2007 Mar;21(3):472-9. doi: 10.1038/sj.leu.2404522. Epub 2007 Jan 11. PMID 17215853
- [Background] Kong Y, Zhang J, Claxton DF, Ehmann WC, Rybka WB, Zhu L, Zeng H, Schell TD, Zheng H. PD-1(hi)TIM-3(+) T cells associate with and predict leukemia relapse in AML patients post allogeneic stem cell transplantation. Blood Cancer J. 2015 Jul 31;5(7):e330. doi: 10.1038/bcj.2015.58. PMID 26230954